CLINICAL TRIAL: NCT00717444
Title: Healthy Activities for Prize Incentives
Acronym: HAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 08-251-2; 1R01DA022739-01A2 (NIH)
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Substance Abuse; HIV Infections
Keywords: Substance Abuse; HIV; Contingency Management; Physical Activity
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): contingency management for abstinence plus 12-step facilitation therapy and contingency management for completing healthy activities
  Interventions: Behavioral: contingency management
- 2 (Experimental): contingency management for abstinence plus 12-step facilitation therapy
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — contingency management for abstinence plus 12-step facilitation therapy
  prizes awarded for target behaviors
  Arms: 2
Behavioral: contingency management — contingency management for abstinence plus 12-step facilitation therapy and contingency management for completing healthy activities
  prizes awarded for target behaviors
  Arms: 1

SUMMARY:
In this Stage 1 therapy development project, we plan to develop, formalize, and derive effect size estimates of a contingency management (CM) therapy that focuses on improving health, especially as related to increasing low intensity physical activities, such as walking, resistance training, and stretching. The Healthy Activities for Prize Incentives (HAPI) intervention will be targeted toward and tested within HIV-positive substance abusers who attend HIV drop-in centers. After initial therapy development in a Stage 1a pilot project with 9 patients, the therapy manuals and materials will be adapted and refined. In a Stage 1b controlled trial, we will recruit and randomize 70 substance abusing HIV-positive patients to (a) HAPI plus 12-step facilitation therapy or (b) contingency management for abstinence plus 12-step facilitation therapy. Each intervention will consist of one weekly individual therapy session for 16 weeks. All participants will provide urine and breath specimens twice weekly that will be tested for opioids, cocaine, methamphetamine, marijuana and alcohol. Patients in both conditions will earn the chance to win prizes for submitting drug-negative specimens, and those randomized to the HAPI condition will also earn the chance to win prizes for engaging in healthy activities. Physical activity levels, drug use, psychological symptoms, and subjective and objective indicators of health (body mass index, waist circumference, blood pressure, viral load) will be measured pre-treatment and at months 2 and 4 (post-treatment), as well as at a 7-month (3 months after treatment) follow-up evaluation. Compared to those receiving 12-step facilitation with contingency management for abstinence, we expect that those in the HAPI condition will participate in more physical activities, decrease drug use to a greater extent, evidence reduced depression, and show trends toward improvements in health indices. If effect sizes in at least the small to medium range are noted across all domains, we will consider the therapy appropriate for further evaluation in a Stage 2 therapy development study.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ and a member of Connections
* Age 18-65 years
* English speaking
* Past-year DSM-IV diagnosis of opioid, cocaine, methamphetamine, alcohol, or marijuana abuse or dependence
* Written permission from one's primary care or infectious disease physician to participate in the study and an exercise program
* Plans to reside in the local area for the next 8 months and
* Willing to sign informed consent

Exclusion Criteria:

* Inability to comprehend the study as assessed by the Informed Consent Quiz and Mini-Mental Status Exam (MMSE)
* Severely disruptive behavior
* In recovery for pathological gambling (due to potential similarity between the contingency management procedure and gambling)
* Serious uncontrolled psychiatric disorder other than substance use disorders that require inpatient hospitalization (e.g., active bipolar disorder, psychosis, suicidal)
* History of myocardial infarction, stroke, unstable angina, coronary artery bypass grafting, angioplasty/stent, uncontrolled arrhythmia, or hyperthyroidism in the past 6 months as reported by patient or physician
* Blood pressure >165/95 mmHg and
* Grossly abnormal findings on indices of physical functioning (>2 SDs above means for sedentary age/gender norms according to ACSM, 2006)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
drug use | baseline and each follow-up

SECONDARY OUTCOMES:
physical activity | baseline and each follow-up
psychological symptoms | baseline and each follow-up
medical outcomes | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- Connections, Inc., Hartford, Connecticut, United States